CLINICAL TRIAL: NCT00158587
Title: A Placebo Controlled, Randomised Evaluation of an Eight Week Primaquine Regimen for the Treatment of Vivax Malaria.
Brief Title: Eight Week Primaquine Regimen for the Treatment of Vivax Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: HealthNet TPO (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIF23
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria; Vivax Malaria
Keywords: Vivax; Treatment; Primaquine; Asia
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: primaquine

SUMMARY:
Plasmodium vivax represents a major health problem throughout the tropics. Outside Africa it accounts for over 50% of cases, affecting an estimated 70-80 million people per year. A substantial proportion of clinical cases are not caused by infective bites of Anopheles spp, but by activation of latent hypnozoites in the liver. These relapses may significantly impede development since each illness may result in 5-15 days of absence from work or school.

Primaquine(PQ) is the only drug available that eliminates hypnozoites, though its use is beset by clinical problems; it may precipitate haemolytic anaemia in individuals deficient in the blood enzyme glucose 6 phosphate dehydrogenase (G6PD). Without affordable G6PD testing, primaquine use is precluded. Evidence suggests, however, that a course of 8 weekly doses may be a safe and effective alternative to the traditional 14 day course of the drug. The aim of the proposed study, therefore, is to test whether 8 weekly doses of primaquine is as effective as the 14 day course at preventing relapse malaria, without the risk of hemolysis in G6PD deficient individuals.

DETAILED DESCRIPTION:
Old evidence suggests that successful PQ therapy is not a function of the length of the course of treatment, nor the circulating concentration of the drug, but of the total dosage administered. The same dose administered over 7 days, 14 days, and 8 weeks equally prevented relapse in vivax malaria. The hemolysis seen in shorter courses is often self-limiting, suggesting that feedback mechanisms up-regulate production of red cells in response to haemolytic challenge. The proposed extended course is likely to be well tolerated in G6PD deficient individuals as a result of these safeguards, especially in this population which has been exposed to the 5 day PQ regimen for a number of years without reported adverse effects.

The aim of the study, therefore, is to test whether an 8 week regimen proves effective, without the associated risk of haemolysis in G6PD deficient individuals. However, operational concerns remain about adherence to this protracted treatment regimen. Therefore we will compare the 8 week course in 2 different groups; the first to be directly observed dosing, the second to be unsupervised dosing using pre-packaged, foil wrapped PQ in appropriately labelled individual boxes, supplied with strong health education messages. This would be appropriate for deployment in a resource-poor setting if it proved effective and safe.

Objectives:

To evaluate whether an eight week primaquine regimen, using single weekly doses, can provide adequate radical cure of vivax malaria under experimental and operational conditions and is safe in and acceptable to a population with glucose 6 phosphate dehydrogenase deficiency. The specific objectives of the study are set out below.

1. Determine the efficacy of an eight-week primaquine regime, using single weekly doses, in preventing relapses of P. vivax infections following supervised versus unsupervised administration of the drug.
2. Compare the efficacy and operational aspects (e.g. adherence) between the two week, eight week supervised and eight week blister package regimes.
3. Monitoring of the effect of 8 week PQ on G6PD deficient individuals.
4. Examine the user acceptability and economic advantages of this course of treatment.

Study population:

Vivax positive individuals from Adizai and Baghicha refugee camps, Pakistan, and Jalalabad, Afghanistan.

Laboratory Examination:

All suspected malaria cases attending basic health units will have thick and thin blood films taken and examined by conventional light microscopy. Cases diagnosed with P. vivax infection will be asked to participate in the study unless the exclusion criteria are met. All patients will then be tested for G6PD deficiency by near patient testing. The test is a colorimetric qualitative test for G6PD in red cells requiring 0.05 ml of blood. In addition, a filter paper blood spot will be collected to allow molecular typing of the parasite. This will differentiate between a new and a relapse infection.

Design

Randomised placebo controlled study comparing the following four study groups:

1. Initial 3 day chloroquine with supervised weekly placebo for 8 weeks.
2. Initial 3 day chloroquine followed by supervised 14 day primaquine treatment.
3. Initial 3 day chloroquine followed by supervised 8 week primaquine treatment (45 mg / week).

All patients will be given health education messages and strongly advised to complete the course. In addition a safety arm will be used for G6PD deficient patients; this will be used to compare PCV with group 3 (above). This will be an 8 week regimen, administered by direct observation, and will receive close monitoring for haemolysis.

Treatment:

All patients will be given a full therapeutic course of chloroquine. Primaquine will be administered to the study groups according to the respective protocol schedule. All relapses and new cases will be re-treated using the same regime and procedure as at the time of admission.

Monitoring:

Patients in treatment groups 1, 2, and 3 will be monitored for the initial 8 weeks of treatment for adverse events; G6PD deficient patients will be monitored for signs of hemolysis every other day for the first 2 weeks of treatment and then once per week (prior to dosing) until completion of the course. Following the treatment period, patients will be monitored for 1 year for the following outcomes:

Primary Efficacy Variable: Proportion with relapse(s) of P. vivax in 12 months of follow-up.

Secondary Efficacy Variables: Time to subsequent relapse episode, number of relapse episodes in 12 months, side effects / adverse events

Patients will be advised to return to the BHU in the event of recurrent symptoms within 12 months following enrolment to the study. A patient will be deemed to have completed the study after 12 months of follow-up. In any event each patient will be contacted once every 2 weeks during the follow-up period in order to collect relevant information. At each episode, a sample of blood will allow molecular typing of the parasite and define whether the patient has a new infection or a relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with P. vivax parasitaemia
* Patients over 3 years
* Patients with G6PD deficiency to a safety trial
* Patients without G6PD deficiency to all other groups.

Exclusion Criteria:

* Children under the age of three
* Pregnant / breast feeding women
* Patients with severe clinical anaemia [Hb<7g/dl]
* Patients with P. falciparum
* Patients unavailable for the duration of study.
* Patients who have taken antimalarial drugs in the 2 weeks prior to consultation.
* Patients with concomitant infections or whose general health is considered too poor.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Variable: Proportion with relapse(s) of P. vivax in 12 months of follow-up. | 2004-March 2007

SECONDARY OUTCOMES:
Secondary Efficacy Variables: Time to subsequent relapse episode | 2004-March 2007
Number of relapse episodes in 12 months | 2004-March 2007
Side effects / adverse events | 2004-March 2007

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rowland, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Leslie T, Mayan I, Mohammed N, Erasmus P, Kolaczinski J, Whitty CJ, Rowland M. A randomised trial of an eight-week, once weekly primaquine regimen to prevent relapse of plasmodium vivax in Northwest Frontier Province, Pakistan. PLoS One. 2008 Aug 6;3(8):e2861. doi: 10.1371/journal.pone.0002861. PMID 18682739